CLINICAL TRIAL: NCT04566107
Title: Self-Management Interventions Using Mobile Health for the Multimorbid
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska (Other)
Collaborators: Greater Plains Collaborative Clinical Data Research Network (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 0445-18-EP
Record Dates: First submitted 2020-05-04; First posted 2020-09-28 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Multiple Chronic Conditions
Keywords: multiple chronic conditions; mobile health; multimorbidity
MeSH Terms: conditions — Multiple Chronic Conditions | interventions — Telemedicine

STUDY DESIGN:
Masking Description: No masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Enhanced Usual Care (No Intervention): The enhanced usual care group will receive evidence-based standardized disease-specific education based on discharge protocols. In addition, individuals in the enhanced usual care group will receive the mobile health platform to record medications taken and BlueTooth devices to record physiologic measurements.
- mHealth (Experimental): The mHealth group will receive evidence-based standardized disease-specific education based on discharge protocols. In addition, the mHealth group will receive the mobile health platform with reminders to take medications and engage in an educational tip. Subjects receive BlueTooth devices to record physiologic measurements.
  Interventions: Behavioral: mHealth intervention
- mHealth Plus (Experimental): The mHealth group plus will receive evidence-based standardized disease-specific education based on discharge protocols. In addition, the mHealth plus group will receive the mobile health platform with reminders to take medications and engage in an educational tip. Participants receive BlueTooth devices to record physiologic measurements. The m-Health Plus group will receive real-time virtual visits with a nurse practitioner/community health worker team. Virtual visits are similar to an office follow-up visit with an health care provider using Zoom technology to allow for face-to-face interaction with the patient.
  Interventions: Behavioral: mHealth Plus

INTERVENTIONS:
Behavioral: mHealth intervention — The intervention promotes self-management and adherence to treatment regimens in patients with multimorbidity. This 8-week SM intervention uses mobile health (m-Health) technology for daily messages and reminders to promote self-monitoring activities. Bluetooth devices provided will depend on the participant's need for self-management; heart failure (scale), diabetes (glucometer), COPD (pulse oximeter) or hypertension (BP machine).
  Arms: mHealth
Behavioral: mHealth Plus — The intervention promotes self-management and adherence to treatment regimens in patients with multimorbidity. This 8-week SM intervention uses tailored self-management strategies (action planning, goal setting, and individual identified support needs) and mobile health (m-Health) technology for virtual visits, daily messages, and self-monitoring activities. The investigators will test the additive impact of having the nurse practitioner/community health worker (NP/CHW) team with the m-health platform. The NP will evaluate physiological and psychosocial status while the CHW will assist in recognizing possible solutions to challenging social determinants of health by identifying community resources and guidance in overcoming barriers. Bluetooth devices provided will depend on the participant's need for self-management; heart failure (scale), diabetes (glucometer), COPD (pulse oximeter) or hypertension (BP machine). Participants will receive reminders through the platform.
  Arms: mHealth Plus

SUMMARY:
The purpose of this pilot study is to evaluate the feasibility and impact of delivering mobile health self-management interventions to improve adherence to the prescribed treatment in a multimorbid population returning home after hospital discharge.

DETAILED DESCRIPTION:
The purpose of this three-group repeated-measures randomized controlled trial is to evaluate the use of mobile health (mHealth) self-management technology as a model of care for individuals with multimorbidity. Specifically, this 8-week self-management intervention uses tailored self-management strategies (action planning, goal setting, and individually identified support needs) and mHealth technology for real-time virtual visits, daily messages, and self-monitoring activities. The investigators are testing the additive impact of having the nurse practitioner/community health worker (NP/CHW) team with the mHealth platform (mHealth Plus). The NP evaluates physiological status by evaluating symptoms and tailoring the intervention specific to the individual's multimorbidity while the CHW will assist in recognizing possible solutions to challenging social determinants of health by identifying community resources and guidance in overcoming barriers.

The following specific aims will be addressed:

Aim 1: To evaluate the feasibility of implementing comparative SM interventions (mHealth and mHealth plus virtual visits with a nurse practitioner and community health worker team) in multimorbid individuals by assessing: a) acceptability of each intervention; b) enrollment (recruitment efficiency, attrition, problems and solutions); c) intervention fidelity (delivery, receipt, enactment of the intervention [benefits and barriers]); and d) data collection (technological transfer of data, instrument reliability, the time required, missing data).

Aim 2: To examine the impact of delivering the m-Health and m-Health plus interventions compared to standard care (SC) in multimorbid individuals on: a) primary outcome: adherence to disease-specific lifestyle behaviors (e.g. diet and medication, and self-monitoring of physiological measures as needed (e.g. weight blood pressure, blood glucose, oxygen saturation); b) secondary outcomes: health related quality of life; c) patient-reported health status; d) symptom status; and e) healthcare utilization.

ELIGIBILITY:
Inclusion Criteria:

1. multimorbid patients with one of 4 chronic conditions (HF, COPD, diabetes or hypertension) and have at least one other chronic disease (i.e., hypertension, cancer, stroke, heart disease, diabetes, arthritis, hepatitis, current asthma, kidney failure, or COPD),
2. adult patients (age 19 and older)
3. access to smart technology (phone or iPad) and internet access or a phone plan large enough for daily interactions; and d) able to hear, speak and read English.

Exclusion Criteria:

1. major surgery while admitted;
2. discharged to somewhere other than home (e.g., long term care facility);
3. receiving home health services;
4. documented dementia; and
5. life expectancy <6 months.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2019-10-14 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Usability and acceptability of the self-management interventions by administering a Usability and Acceptability tool | 60 days after enrolled
  A Usability and Acceptability investigator developed tool.
Enrollment of participants to the comparative self-management (SM) interventions by calculating frequency and percentage of available participants and enrolled participants. | 90 days after enrolled
  measure of enrollment and recruitment
Number of times the participant records activities within the application. | 90 days after enrollment
  Measurement of engagement with the application, participant records will be downloaded from the application and frequency and percent will be calculated

SECONDARY OUTCOMES:
Frequency and percent of the participants recording a weight in pounds in the mHealth app | 30 days after intervention initiated
  monitoring of physiological measures for each of the physiologic parameters appropriate for the participants chronic disease (number of weights recorded for heart failure participant)
Frequency and percent of the participants recording a weight in pounds in the mHealth app | 60 days after intervention initiated
  monitoring of physiological measures for each of the physiologic parameters appropriate for the participants chronic disease (number of weights recorded for heart failure participant)
Frequency and percent of the participants recording a weight in pounds in the mHealth app | 90 days after intervention initiated
  monitoring of physiological measures for each of the physiologic parameters appropriate for the participants chronic disease (number of weights recorded for heart failure participant)
Frequency and percent of the participants recording a blood pressure (BP) in the mHealth app | 30 days after intervention initiated
  monitoring of physiological measures for each of the physiologic parameters appropriate for the participants chronic disease (number of BP recorded for hypertension participant)
Frequency and percent of the participants recording a blood pressure (BP) in the mHealth app | 60 days after intervention initiated
  monitoring of physiological measures for each of the physiologic parameters appropriate for the participants chronic disease (number of BP recorded for hypertension participant)
Frequency and percent of the participants recording a blood pressure (BP) in the mHealth app | 90 days after intervention initiated
  monitoring of physiological measures for each of the physiologic parameters appropriate for the participants chronic disease (number of BP recorded for hypertension participant)
Frequency and percent of the participants recording a pulse oximetry in the mHealth app | 30 days after intervention initiated
  monitoring of physiological measures for each of the physiologic parameters appropriate for the participants chronic disease. (number of oximetry readings recorded for chronic obstructive pulmonary disease (COPD) participant)
Frequency and percent of the participants recording a pulse oximetry in the mHealth app | 60 days after intervention initiated
  monitoring of physiological measures for each of the physiologic parameters appropriate for the participants chronic disease (number of oximetry readings recorded for (COPD) participant)
Frequency and percent of the participants recording a pulse oximetry in the mHealth app | 90 days after intervention initiated
  monitoring of physiological measures for each of the physiologic parameters appropriate for the participants chronic disease (number of oximetry readings recorded for the chronic obstructive pulmonary disease (COPD) participant)
Frequency and percent of the participants recording a blood glucose in the mHealth app | 30 days after intervention initiated
  monitoring of physiological measures for each of the physiologic parameters appropriate for the participants chronic disease (number of blood glucose readings recorded for the diabetic participant)
Frequency and percent of the participants recording a blood glucose in the mHealth app | 60 days after intervention initiated
  monitoring of physiological measures for each of the physiologic parameters appropriate for the participants chronic disease (number of blood glucose readings recorded for the diabetic participant)
Frequency and percent of the participants recording a blood glucose in the mHealth app | 90 days after intervention initiated
  monitoring of physiological measures for each of the physiologic parameters appropriate for the participants chronic disease (number of blood glucose readings recorded for the diabetic participant)
Health related quality of life assessed by the EQ-5D-5L developed by the EuroQol group scored as an index and a visual analogue scale. | 30 days after intervention initiated
  monitoring of physiological measures for each of the physiologic parameters appropriate for the participants chronic disease (number of blood glucose readings recorded for the diabetic participant)
Health related quality of life assessed by the EQ-5D-5L developed by the EuroQol group scored as an index and a visual analogue scale. | 60 days after intervention initiated
  Measure of quality of life
Health related quality of life assessed by the EQ-5D-5L developed by the EuroQol group scored as an index and a visual analogue scale. | 90 days after intervention initiated
  measure of quality of life
Patient Reported Outcomes Measurement Information System (PROMIS®) (Promis29 V2.0) score of mobility, self-care, usual activities, pain/ discomfort, anxiety/ depression and a visual analogue scale rating of health today | 30 days after intervention initiated
  Measure of health status and symptoms
Patient Reported Outcomes Measurement Information System PROMIS® (Promis29 V2.0) score of mobility, self-care, usual activities, pain/ discomfort, anxiety/ depression and a visual analogue scale rating of health today | 60 days after intervention initiated
  measure of health status and symptoms
Patient Reported Outcomes Measurement Information System PROMIS® (Promis29 V2.0) score of mobility, self-care, usual activities, pain/ discomfort, anxiety/ depression and a visual analogue scale rating of health today | 90 days after intervention initiated
  measure of health status and symptoms
Emergency rooms visits and re-hospitalizations assessed by frequency and percent assessed by reviewing the electronic medical record | 30 days after intervention initiated
  measure of health care utilization
Emergency rooms visits and re-hospitalizations assessed by frequency and percent assessed by reviewing the electronic medical record | 60 days after intervention initiated
  measure of health care utilization
Emergency rooms visits and re-hospitalizations assessed by frequency and percent assessed by reviewing the electronic medical record | 90 days after intervention initiated
  measure of health care utilization

CONTACTS AND LOCATIONS:
Overall Officials: Myra S Schmaderer, PhD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, College of Nursing, Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No